CLINICAL TRIAL: NCT01868828
Title: A Multicenter, Double Arms, Prospective Phase 4 Study to Evaluating the Efficacy and Safety of Combination Therapy of PAD Versus VCD Treatment in Previously Untreated Subjects With Multiple Myeloma.
Brief Title: A Study of PAD Versus Velcade, Cyclophosphamide and Dexamethasone (VCD) Treatment in Subjects With Multiple Myeloma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jin Lu, Associate Chief Physician, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAD VS VCD Clinical Protocol
Record Dates: First submitted 2013-05-22; First posted 2013-06-05 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Combination Therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PAD Followed by ASCT (Experimental): Drug: Bortezomib(1.3mg/m2, iv, on day 1, 4, 8, 11)
  Drug: Epidoxorubicin(15 mg/m2, iv, on days 1-4)
  Drug: Dexamethasone(40mg, orally, on days 1-4)
  After received induction therapy, patients will proceed to receive ASCT based on the willing of the patients and the decision of the investigators.
  Not suitable for transplant patients will continue accept treatment for 8 cycles.
  Interventions: Drug: PAD; Other: ASCT
- VCD Followed by ASCT (Experimental): Drug: Bortezomib (1.3mg/m2, iv, on day 1, 4, 8, 11)
  Drug: Cyclophosphamide (200mg/m2, orally, on days 1-5)
  Drug: Dexamethasone(40mg, orally, on days 1-4)
  After received induction therapy, patients will proceed to receive ASCT based on the willing of the patients and the decision of the investigators.
  Not suitable for transplant patients will continue accept treatment for 8 cycles.
  Interventions: Drug: VCD; Other: ASCT

INTERVENTIONS:
Drug: PAD — Induction Therapy of PAD for 4 cycles.
  Other Names: Induction Therapy
  Arms: PAD Followed by ASCT
Drug: VCD — Induction Therapy of VCD for 4 cycles.
  Other Names: Induction Therapy
  Arms: VCD Followed by ASCT
Other: ASCT — Not suitable for transplant patients will continue accept treatment for 8 cycles.

SUMMARY:
A multicenter, double arms, prospective randomized controlled phase 4 study. Approximately 50 previously untreated subjects with multiple myeloma will be enrolled. The study will consist of 6 phases, screening, treatment and follow-up.

DETAILED DESCRIPTION:
Screening

At the screening visit, informed consent will be obtained from all subjects who are deemed potentially eligible for enrollment in the study, according to the protocol-specified inclusion and exclusion criteria.

Treatment

Eligible patients are randomly assigned to receive either treatment PAD or VCD. All eligible subjects will be evaluated after 4 cycles treatment. According to the assessment of researchers and the willingness of patients to decide whether to autologous stem-cell transplantation (ASCT). Suitable for transplant patients will accept hematopoietic stem cell transplantation. Not suitable for transplant patients will continue accept treatment for 8 cycles. The patients who accept more than 4 cycles treatment will receive efficacy evaluation.

Follow-up

All patients will receive 12 months of follow-up after the treatment period. Follow-up at 4, 6, 8 and 12 month after the treatment period respectively. Subjects who have disease progression or accept other resistance myeloma therapy during the 12 months of follow-up phase will stop assessed about the study and start followed up only for survival status every 6 months through telephone interviews or to research center follow-up. All patients will accept the follow-up for survival until last case patient who complete follow-up.

Safety will be evaluated throughout the study by assessment of adverse events (AEs), physical examination, vital signs and clinical laboratory findings.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged <65 years.
2. Previously untreated subjects with multiple myeloma.
3. No clinically significant cardiac amyloidosis (Echocardiography septal≤10mm, brain natriuretic peptide (BNP) < 500).
4. Pulmonary infection (if any) must be controlled effectively.
5. Chronic viral hepatitis (if any) must be controlled effectively.(Subjects with HBs Ag positive need to monitor hepatitis B virus-DNA (HBV-DNA )quantitative test regularly）；
6. Liver function (aminotransferase, bilirubin）?2 x the upper limit of normal (ULN).
7. Expected lifetime More than 3 months.
8. Be able to read and sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

1. Patients with relapsed multiple myeloma.
2. Need to change the program according to the researchers' evaluated patients with disease progression during treatment.
3. Had uncontrolled or severe cardiovascular disease. Had a myocardial infarction within 6 months of enrolment, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, clinically significant pericardial disease, or cardiac amyloidosis.
4. Has a history of allergic reaction to compounds containing boron or mannitol.
5. Severe neuropathy may affect the treatment, according to the researchers to determine.
6. According to the program or the investigator's judgment, the patient is suffering from a serious physical illness or mental illness may interfere with participation in this clinical study.
7. Concurrent treatment with another investigational agent.
8. Pregnant or breast-feeding women.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate | Up to cycle 4 (with 28 days per cycle).

SECONDARY OUTCOMES:
Safety | At baseline, on day 1 of each cycle, and after 4, 6, 12 and 18 months of follow-up.
  Safety evaluations will be based on scheduled clinical laboratory tests, electrocardiogram or cardiac ultrasonography (when appropriate), vital signs, physical examination and number of adverse events.
Overall Response Rate | At baseline, on day 28 of each cycle for 4 cycles.
  Overall response rate included Complete Response (CR), Very good partial response (VGPR) and PR, before the new treatment, two consecutive evaluations are in line with defined criteria in order to confirm the efficacy evaluation.
Time To Response | At baseline, on day 28 of each cycle for 4 cycles.
1-year Survival Rate | At baseline, on day 28 of each cycle, and after 4, 6, 12 and 18 months of follow-up.
Overall Survival | At baseline, on day 28 of each cycle, and after 4, 6, 12 and 18 months of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Lu, PhD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Institute of Hematology, Peking University, Beijing, Beijing Municipality, China